CLINICAL TRIAL: NCT05373017
Title: Delirium and Neuropsychological Recovery Among Emergency General Surgery Survivors (DANE)
Brief Title: Delirium and Neuropsychological Recovery Among Emergency General Surgery Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Indiana University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0545; A539714 (Other: UW Madison); Protocol Version 4/20/2025 (Other: UW Madison); SMPH/SURGERY/TRAUMA (Other: UW Madison); 1R01AG076489-01 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DANE Recovery Model (Experimental): The delivery of the model will occur in five phases that correspond to the known stages of recovery after surgery. During the acute stage (0 - 1 month after surgery), participants will undergo the initial case review and two initial virtual visits, and the development of the recovery care plan. During the recovery (2 - 6 months after surgery) and maintenance (7-12 months after surgery) stages, the participants will undergo the interaction phase of the DANE Recovery Model.
  Interventions: Other: DANE Recovery Program
- Usual Care (Other): Participants will receive the usual rehabilitation and post-operative care.
  Interventions: Other: DANE Recovery Program; Other: Questionnaires

INTERVENTIONS:
Other: DANE Recovery Program — Virtual visits with care coordinator to carry out an individualized recovery plan
Other: Questionnaires — Physical, cognitive, and psychological assessments
  Arms: Usual Care

SUMMARY:
This study will evaluate the usefulness of the Urgent and Emergency Surgery (UES) Delirium Recovery Model. It is hypothesized that the cognitive, physical and psychological recovery of older UES delirium survivors will be improved through the use of the DANE Recovery Model. Participants can expect to be on the study for 18 months.

DETAILED DESCRIPTION:
This is a multi-site, two-arm, single-blinded randomized controlled clinical trial to evaluate the efficacy of the DANE Recovery Model to improve the cognitive, physical and psychological recovery of older UES delirium survivors. At or near the time of discharge, enrolled participants will be randomized to receive the DANE Recovery Model or usual care. The hypothesis is that, after 18 months, older UES delirium survivors who are randomized to the DANE Recovery Model will experience more favorable cognitive, physical and psychological recovery in comparison to those randomized to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 65 years and older
* Admitted to one of the participating hospitals
* Undergone an abdominal orthopedic, skin, or vascular surgery in an emergency or unplanned fashion
* English-speaking
* Able to provide consent or have a legally authorized representative to provide consent
* Access to a telephone or an internet connected computer or smart device
* Discharged to home or sub-acute rehabilitation
* At least one episode of delirium or subsyndromal delirium, i.e. screen positive on at least one out of the four items on the Confusion Assessment Method-ICU (CAM-ICU) in the period prior to discharge from acute care.

Exclusion Criteria:

* A self-reported diagnosis of cancer with short life expectancy
* A history of dementing illnesses and other neurodegenerative disease such as Alzheimer's disease (AD), Parkinson disease, or vascular dementia, or current prescription of anti-dementia medication, or ruled out by Functional Activities Questionnaire (FAQ) score defining dementia; a history of significant traumatic brain injury
* Acute or subacute neurologic deficit expected to prevent independent living after hospital discharge, e.g., a history of a significant traumatic brain injury
* Have any spinal cord injury with persistent neurologic deficit at the time of study enrollment
* Incarcerated or homeless at the time of study enrollment
* Acquired neurologic injury (stroke, traumatic brain injury, cerebral edema/swelling, anoxic brain injury, or any other acute/subacute severe neurologic deficit) as the admitting diagnosis or a new event during the course of hospitalization (confirmed by EMR)
* A history of bipolar disorder or schizophrenia (confirmed by EMR)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in overall cognitive recovery | Baseline, 6 months, 12 months, and 18 months
  Change in score on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) cognitive screening assessment. The measure consists of 12 subtests that contribute to a total score and Index scores across five domains: Immediate Memory, Visuospatial-Constructional, Language, Attention, and Delayed Memory. Index scores are converted to age-based standard scores (Mean = 100, Standard Deviation = 15)

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, 6 months, 12 months, and 18 months
  Change in overall physical recovery will be assessed using Short Physical Performance Battery (SPPB). SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests, and yields a performance score of 0-12; 0-4 poor, 5-7 intermediate, 8-12 good.
Change in overall physical recovery | Baseline, 6 months, 12 months, and 18 months
  Change in overall physical recovery will be assessed using 36-Item Short Form Survey (SF-36). SF-36 scale has eight components (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health).
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 6 months, 12 months, and 18 months
  Change in overall psychological recovery will be assessed using Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a nine-item depression scale with a total score from 0 to 27, with higher scores indicating greater depression.
General Anxiety Disorder-7 (GAD-7) . | Baseline, 6 months, 12 months, and 18 months
  Change in overall psychological recovery will be assessed using General Anxiety Disorder-7 (GAD-7) to determine the impact of the intervention on participant's mood and anxiety. The GAD-7 is a seven-item anxiety scale with a total score from 0 to 27, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Zarzaur, MD, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - SwedishAmerican Hospital, Rockford, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Wisconsin, Madison, Wisconsin
  - Meriter Hospital, Madison, Wisconsin
  - East Madison Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gardner L, Bylund P, Robbins S, Holler E, Shojaei F, Shojaei F, Seidman M, Holden RJ, Fowler NR, Zarzaur B, Barboi C, Boustani M. Agile monitoring dashboard for clinical research studies. Trials. 2024 Nov 29;25(1):802. doi: 10.1186/s13063-024-08646-0. PMID 39609928
- [Derived] Mohanty S, Holler E, Ortiz D, Meagher A, Perkins A, Bylund P, Khan B, Unverzagt F, Xu H, Ingraham A, Boustani M, Zarzaur B. Delirium and neuropsychological recovery among emergency general surgery survivors (DANE): study protocol for a randomized controlled trial and collaborative care intervention. Trials. 2023 Oct 3;24(1):634. doi: 10.1186/s13063-023-07670-w. PMID 37789461
- [Derived] Mohanty S, Holler E, Ortiz D, Meagher A, Perkins A, Bylund P, Khan B, Unverzagt F, Xu H, Ingraham A, Boustani M, Zarzaur B. Delirium and Neuropsychological Recovery among Emergency General Surgery Survivors (DANE): study protocol for a randomized controlled trial and collaborative care intervention. Res Sq [Preprint]. 2023 Sep 7:rs.3.rs-3185716. doi: 10.21203/rs.3.rs-3185716/v1. PMID 37720054